CLINICAL TRIAL: NCT04697108
Title: Reliability of a Proprioception Teste in Swimmers Athletes
Brief Title: Reliability of a Proprioception Test in Swimmers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: São Paulo State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FIS190111
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Athletes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proprioception Test (TRMOPL) (Other): In the Familiarization stage (1), the TRMOPL was applied by means of a single evaluator with the aim of knowledge and understanding of the test. After five minutes, step (2) test started. In this step, the test was applied twice, by different evaluators, with an interval of five minutes between applications (inter-rater reliability). Ten minutes after the end of the tests, step (3) retest (intra-rater reliability) was started, following the same procedures as in step 2. The order of the evaluators was randomized through a draw in Excel, the order of randomization of the steps (2) and (3) was the same in order not to influence intra-rater reliability.
  Interventions: Other: Shoulder reproduction teste assisted by laser pointer

INTERVENTIONS:
Other: Shoulder reproduction teste assisted by laser pointer — In the step (1) of Familiarization in which the SRTLP was applied through a single evaluator with the aim of knowledge and understanding of the test. After five minutes, step (2) test started. In this step, the test was applied twice, by different evaluators, with an interval of five minutes between applications (inter-rater reliability). Ten minutes after the end of the tests, step (3) retest (intra-rater reliability) was started, following the same procedures as in step 2. The order of the evaluators was randomized through a draw in Excel, the order of randomization of the steps (2) and (3) was the same in order not to influence intra-rater reliability

SUMMARY:
To evaluate the intra- and inter-rater reliability of a test of active shoulder proprioception with a laser pointer in swimming athletes and to describe the profile of the proprioception measures characterizing the sample according to the specialty within the sport and the category of the athletes.

DETAILED DESCRIPTION:
Introduction: Obtaining the reliability of an evaluative instrument is of paramount importance for its applicability in the field of clinical physiotherapy and in the sports field, providing consistent and real measures. Shoulder proprioception assessments have started to appear on the scientific scene in recent years and several tools, methods and protocols are being studied. However, the lack of standardization of protocols and application in different populations produces inconsistencies in the findings, thus hindering the use of these models. Thus, standardizing the application of the test and investigating a population different from what appears in the scientific scenario in relation to sports, such as swimming athletes, seems to be relevant and would contribute to the use of scientific evaluative models in the clinical environment. Objectives: To evaluate the intra- and inter-rater reliability of a test of active shoulder proprioception with a laser pointer in swimming athletes and to describe the profile of the proprioception measures characterizing the sample according to the specialty within the sport and the category of the athletes. Methods: Study of intra- and inter-rater reliability of the shoulder proprioception test with a laser pointer, composed of 48 young male and female swimming athletes, aged between 12 and 20 years. It will be carried out in three stages: (1) Familiarization, (2) Test and (3) Retest, all stages will take place on the same day, and stages 2 and 3 will be performed by two different evaluators. To characterize the sample, descriptive statistics will be used by means of central tendency and variability, for all variables collected. Relative reliability will be tested by the Intraclass Correlation Coefficient (ICC), with a 95% confidence interval. The ICC will be interpreted as values <0.5 indicate low reliability, between 0.5 and 0.75, moderate reliability, between 0.75 and 0.9, good reliability and values> 0.90 excellent reliability. And the absolute reliability will be verified by means of the standard error of the measurement (EPM), by values of minimum detectable change (MMD), and the coefficient of variation (CV).

ELIGIBILITY:
Inclusion Criteria:

* Male and female swimming athletes;
* Between 12 and 26 years old;
* Train regularly and be members of swimming teams in the 4th Region of the State of São Paulo, and athletes from the São Paulo Aquatic Federation (FAP),
* Reporting the absence of anemia, inflammatory process, diabetes, cardiovascular disease, episodes of muscle - tendon or osteoarticular injury in the lower, upper and / or spine members in the last three months.

Exclusion Criteria:

* Practice of sports for less than 1 year.
* Use anti-inflammatory and / or analgesic drugs for less than 24 hours before the test.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Joint Position Sense | One hour
  the movement reproduction test was applied by a laser pointer and the measurements presented were angular deviation in degrees.

SECONDARY OUTCOMES:
Shoulder Pain | 5 minutes
  Pain measurements were performed using a visual pain scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo State, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Individual data will not be released, because particpants are under eighteen.